CLINICAL TRIAL: NCT01156337
Title: Sodium Management in Acute and Chronic Phases in Patients With New York Heart Association Class III (Class C) Heart Failure. Short and Long Term Findings.
Brief Title: Sodium Management in Acute and Chronic Heart Failure
Acronym: SMAC-HF
Status: Completed | Type: Observational
Sponsor: Ospedale G. F. Ingrassia (Other)
Collaborators: University of Palermo (Other); University of Naples (Other); Buccheri La Ferla Hospital, Palermo (Other)
Other Study IDs: G.F. Ingrassia Hospital,Italy
Record Dates: First submitted 2010-07-01; First posted 2010-07-02 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2007-08

CONDITIONS: Heart Failure
Keywords: Heart failure III NYHA class; Furosemide; Sodium; water restriction; decompensated heart failure; Hypertonic saline solution; Moderate sodium restriction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- low sodium diet 80 mmol/day
- moderate sodium intake 120 mmol/day

SUMMARY:
The study was aimed to verify the effects of Hypertonic saline solution (HSS) and a moderate sodium (Na) restriction plus high furosemide dose in the short term (hospitalization time) and a moderate Na restriction in the long term on readmissions and mortality in patients in III NYHA class.

ELIGIBILITY:
Inclusion Criteria:

* Decompensated HF due to ischemic or nonischemic cardiomyopathy,
* >18 years of age,
* HF according to Framingham criteria
* NYHA functional class III
* EF <40%,
* Serum creatinine <2,5 mg/dL
* BUN <60 mg/dL,

Exclusion criteria:

* NYHA class > III or < III,
* Cerebral vascular disease,
* Dementia,
* Cancer,
* Uncompensated diabetes,
* Severe hepatic disease
* Patients requiring pacemaker
* Previous RCT implantation
* Alcoholic habit

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients in III NYHA class HF
Sampling Method: Non-Probability Sample
Dates: Start 2000-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
readmission for HF worsening

SECONDARY OUTCOMES:
mortality

CONTACTS AND LOCATIONS:
Locations (1):
- GF Ingrassia Hospital, Palermo, Italy